CLINICAL TRIAL: NCT03042884
Title: Wearable Exercise Trackers in Cancer Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0671
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Benign Neoplasms; In Situ Neoplasms; Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Benign Neoplasms; In Situ Neoplasms; Malignant Neoplasms of Independent (Primary) Multiple Sites; Wearable exercise trackers; Questionnaires; Surveys
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable Exercise Trackers - Inpatient Group (Experimental): Questionnaires completed at baseline and within 24 hours of discharge.
  Participant given a wearable exercise tracker to be worn 24 hours a day while in the acute inpatient rehabilitation unit.
  Interventions: Behavioral: Questionnaires; Device: Wearable Exercise Tracker Watch
- Wearable Exercise Trackers - Outpatient Group (Experimental): Questionnaires completed at baseline and again in 14 days.
  Participant given a wearable exercise tracker to be worn 24 hours a day for 14 days.
  Interventions: Behavioral: Questionnaires; Device: Wearable Exercise Tracker Watch

INTERVENTIONS:
Behavioral: Questionnaires — Inpatient Group: Participants complete a questionnaire about any symptoms they may have had in the past 24 hours. The questionnaire should take about 5 minutes to complete.
  Within 24 hours of being discharged, same questionnaire about symptoms and a questionnaire about experience with the wearable exercise tracker. These questionnaires should take about 10 minutes total to complete.
  Outpatient Group: Participants complete 2 questionnaires about any symptoms they may have had in the past 24 hours and their current level of physical function. These should take about 10 minutes total to complete.
  At the end of the 14-day period, participant called by the study staff to remind them to complete the same 2 questionnaires about symptoms and level of physical function. Participants complete another questionnaire about their experience with the wearable exercise tracker. These questionnaires should take about 15 minutes total to complete.
  Other Names: Surveys
Device: Wearable Exercise Tracker Watch — Inpatient Group: Participants receive a wearable exercise tracker watch upon admission to acute inpatient rehabilitation unit. Participant to wear the exercise tracker watch on their wrist for 24 hours a day. Device to be returned within 24 hours before being discharged.
  Outpatient Group: Participants receive a wearable exercise tracker watch to wear on their wrist for 24 hours a day for 14 days. Device to be returned at next visit.

SUMMARY:
The goal of this research study is to learn how useful a wearable exercise tracker watch is to monitor your physical activity.

This is an investigational study.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Inpatient:

If you agree to take part in this study, you will complete a questionnaire about any symptoms you may have had in the past 24 hours. The questionnaire should take about 5 minutes to complete.

You will receive a wearable exercise tracker watch and an iPod touch. You should wear the exercise tracker watch on your wrist for 24 hours a day (or as much as possible) while you are in the acute inpatient rehabilitation unit, even when you sleep. The iPod touch will be used to sync the data from the tracker watch to the study's activity database so the study team can view your activity. Instructions on how to use the tracker and how to sync the trackers to the iPod touch will be given to you and demonstrated by the research staff.

The research coordinator will be available to help you with any issues you may have while taking part in the study and will call you to answer any questions. You will be called on Day 3 (+/- 2 days) of the study and again at the end of the study. These calls should last about 5 minutes each time.

The wearable tracker will record your steps, sleep time, time spent doing physical activity, heart rate, and distance. You may choose to record the food you eat and mood. Your ability to keep wearing the watch will be measured.

You should wear the band loosely enough that it can move back and forth on your wrist. If it becomes too bothersome, you can take the watch off and put it back on after an hour.

You should regularly clean the band and your wrist, especially after your rehabilitation sessions. Rinse the band with water or wipe it with a small amount of rubbing alcohol. Do not use hand soap, body soap, dish soap, hand sanitizers, cleaning wipes or household cleaners which could get trapped beneath the band and irritate your skin. Always dry the band well before putting it back on.

If any of the devices are lost, stolen, or broken, you should tell the study staff right away. They will be replaced at no cost to you as long as you have followed the study doctor's instructions. After you complete the study, we ask that you return the devices to the study staff.

Within 24 hours before you are discharged, you will return the devices to the research staff. You will be asked to complete the same questionnaire about your symptoms and a questionnaire about your experience with the wearable exercise tracker. These questionnaires should take about 10 minutes total to complete. If you are unable to complete them in person, you will be given the option to complete them over the phone or electronically after you have been discharged. If you choose to complete them electronically, your e-mail address will be collected so the survey link can be sent to you. We ask that you complete the questionnaires within 1 week after you are discharged.

Information will be collected from your medical records about your daily living at the beginning and at the end of the study. Basic information, such as your name, date of birth, race, gender, economic background, and medical record number will also be collected.

Length of Study:

You participation on this study will be over after you complete the second set of questionnaires.

Outpatient:

If you agree to take part in this study, you will complete 2 questionnaires about any symptoms you may have had in the past 24 hours and your current level of physical function. These should take about 10 minutes total to complete.

You will receive a wearable exercise tracker watch and an iPod touch. You should wear the exercise tracker watch on your wrist for 24 hours a day (or as much as possible) while you are in the acute inpatient rehabilitation unit, even when you sleep. The iPod touch will be used to sync the data from the tracker watch to the study's activity database so the study team can view your activity. Instructions on how to use the tracker and how to sync the trackers to the iPod touch will be given to you and demonstrated by the research staff.

The research coordinator will be available to help you with any issues you may have while taking part in the study and will call you to answer any questions. You will be called on Day 3 (+/- 2 days) of the study and again at the end of the study. These calls should last about 5 minutes each time.

The wearable tracker will record your steps, sleep time, time spent doing physical activity, heart rate, and distance. You may choose to record the food you eat and mood. Your ability to keep wearing the watch will be measured. No identifying information will be used on the devices.

You should wear the band loosely enough that it can move back and forth on your wrist. If it becomes too bothersome, you can take the watch off and put it back on after an hour.

You should regularly clean the band and your wrist, especially after your rehabilitation sessions. Rinse the band with water or wipe it with a small amount of rubbing alcohol. Do not use hand soap, body soap, dish soap, hand sanitizers, cleaning wipes or household cleaners which could get trapped beneath the band and irritate your skin. Always dry the band well before putting it back on.

If any of the devices are lost, stolen, or broken, you should tell the study staff right away. They will be replaced at no cost to you as long as you have followed the study doctor's instructions. After you complete the study, we ask that you return the devices to the study staff.

At the end of the 14-day period, you will be called by the study staff to remind you to complete the same 2 questionnaires about your symptoms and level of physical function. You will complete another questionnaire about your experience with the wearable exercise tracker. These questionnaires should take about 15 minutes total to complete.

If you choose to complete these forms electronically, they will be made available online with a link on the iPod. You may also choose to complete the questionnaires over the phone.

You will be asked to return the wearable tracker and iPod Touch to the research coordinator at your next routine clinic visit. If you are unable to return to the clinic, you will be asked to mail back the devices with the FedEx postage paid envelope provided to you when you started the study.

Basic information, such as your name, date of birth, race, gender, economic background, and medical record number will also be collected.

Length of Study:

You participation on this study will be over after you complete the second set of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with literacy as demonstrated by reading and signing informed consent form
2. At least 18 years of age, since the rehabilitation unit and physical medicine and rehabilitation clinic is open to patients 18 years of age or older
3. Patients admitted to the acute inpatient rehabilitation unit and those seen in the Physical Medicine and Rehabilitation outpatient clinic
4. Capable of completing questionnaire in English

Exclusion Criteria:

1) Patients currently using a wearable activity tracker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Usefulness of Exercise Tracker in Acute Inpatient Rehabilitation Unit Per Edmonton Symptom Assessment Scale (ESAS-FS) | 14 days
  Exercise tracker considered useful if at least 2/3 patients consider it as useful.
Usefulness of Exercise Tracker as an Outpatient Per Edmonton Symptom Assessment Scale (ESAS-FS) | 14 days
  Exercise tracker considered useful if at least 2/3 patients consider it as useful.
Usefulness of Exercise Tracker in Acute Inpatient Rehabilitation Unit Per Patient Reported Outcomes Measurement Information System (PROMIS) | 14 days
  Exercise tracker considered useful if at least 2/3 patients consider it as useful.
Usefulness of Exercise Tracker as an Outpatient Per Patient Reported Outcomes Measurement Information System (PROMIS) | 14 days
  Exercise tracker considered useful if at least 2/3 patients consider it as useful.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org